CLINICAL TRIAL: NCT01340131
Title: Open Label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics of Telmisatan 40mg and S-Amlodipine 5mg as a Fixed Dose Combination Tablet Compared With Combination Therapy in Healthy Volunteers
Brief Title: CKD-828 (40/5mg) Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Jin Kim / Director, Clinical Research Department
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 130HPS10G
Record Dates: First submitted 2011-03-30; First posted 2011-04-22 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: CKD-828; Hypertension; Primary Hypertension; Healthy Volunteer; S-Amlodipine; Telmisartan; Amlodipine; Pharmacokinetic; Phase 1
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-828(Fixed Dose Combination) (Experimental): Single oral dose of a FDC tablet consisting of Telmisatan 40mg/S-Amlodipine 5mg Intervention
  Interventions: Drug: CKD-828
- Free combination Therapy (Active Comparator): Co-administration of single oral doses of a 40mg tablet of Telmisatan and a 5 mg tablet of S-Amlodipine
  Interventions: Drug: Combination Therapy

INTERVENTIONS:
Drug: CKD-828 — Drug: Telmisartan 40mg + S-Amlodipine 5mg(FDC) Tablet, Oral, Once Daily
  Arms: CKD-828(Fixed Dose Combination)
Drug: Combination Therapy — Drug: Telmisartan 40mg Tablet, Oral, Once Daily
  Drug: S-amlodipine 5mg Tablet, Oral, Once Daily
  Arms: Free combination Therapy

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics of CKD-828 (Fixed Dose Combination Tablet; Telmisartan and S-Amlodipine) in healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* A healthy volunteer between 20 and 55 years old with body weight within 20% of ideal body weight.
* Have not any congenital or chronic diseases and medical symptom.
* Appropriate for the study judging from examinations(interview, vital signs, 12-lead ECG, physical examination, blood, urinalysis result on screening).
* Able to participate in the entire trial.
* Signed the informed consent form prior to the study participation.

Exclusion Criteria:

* Take metabolic enzyme inducing or inhibiting drugs like barbiturates within 28 days prior to the first IP administraion.
* The evidence of acute disease within 28 days prior to the first IP administraion.
* Disease(ex: imflammatory intestinal disease, gastric or duodenal ulcer ,hepatic diseasehistory , gastro intestinal surgery exept for appendectomy)that may influence on the absorption, distribution, metabolism and excretion of the drug(s).
* Relevant hypersensitivity against drug or clinically significant allergic diseases except mild rhinitis that doesn't need medication.
* Hypersensitivity Telmisartan or Amlodipine.
* SBP<90mmHg or DBP<50mmHg.
* Abnormal laboratory result(s): AST or ALT > 1.25 times of upper limit / Total bilirubin > 1.5 times of upper limit.
* A drug abuse or a heavy caffeine consumer (more than 5 cups per a day) or a heavy smoker(more than 10 cigarettes per a day) or a regular alcohol consumer(more than 30g/day) or drinking within 7days prior to the first IP administration.
* Diet(Especially, grapefruit juice-within 7 days prior to the first IP administraion) that may influence on the absorption, distribution, metabolism and excretion of the drug(s).
* Donated whole blood within 60 days prior to the first IP administraion.
* Participated in the other clinical trials within 90days prior to the first IP administraion.
* Medicine within 10 days prior to the first IP administraion? Does the medication affect this trial.
* Appropriate for the trial judging from principal investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Cmax after administration of CKD-828(Fixed Dose Combination) tablet and co-administration of corresponding dose of Telmisartan and S-Amlodipine as individual tablets. | up to 168 hours postdose
The area under the plasma concentration-time curve (AUC) after administration of CKD-828(Fixed Dose Combination) tablet and co-administration of corresponding dose of Telmisartan and S-Amlodipine as individual tablets. | up to 168 hours postdose

SECONDARY OUTCOMES:
Tmax and t1/2 after administration of CKD-828(Fixed Dose Combination) tablet and co-administration of corresponding dose of Telmisartan and S-Amlodipine as individual tablets. | up to 168 hours postdose
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 22days

CONTACTS AND LOCATIONS:
Overall Officials: Eunyoung Kim, Principal Investigator — Inje University
Locations (1):
- Inje University Pusan Paik Hospital, Pusan, South Korea